CLINICAL TRIAL: NCT01849796
Title: Transcranial Stimulation (TDCS) For The Treatment of Neuropathic Facial Pain.
Acronym: TDCS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigators moved to other institutions
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 148-10
Record Dates: First submitted 2012-12-27; First posted 2013-05-09 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Facial Pain
Keywords: tDCS; Neuropathic; Facial; Pain; Neuralgia; deafferentation; Trigeminal
MeSH Terms: conditions — Facial Pain; Facies; Pain; Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Anodal tDCS (Active Comparator): Group A will receive one block of real excitatory anodal tDCS over the motor cortex and one block of sham.
  Interventions: Device: tDCS
- Arm B: Cathodal tDCS (Sham Comparator): Group B will receive one block of inhibitory cathodal tDCS over the somatosensory cortex and one block of sham.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — TDCS/sham will be delivered using the battery-operated device Phoresor II Auto with two saline-soaked sponge electrodes. To deliver excitatory (anodal) tDCS over the motor cortex, the main electrode will be placed over the motor cortex on the hemisphere contralateral to the major source of pain. The second electrode will be placed on the skin overlying the supraorbital region ipsilateral to the affected area. To deliver inhibitory (cathodal) tDCS, the main electrode will be placed over the somatosensory cortex on the hemisphere contralateral to the major source of pain. The second electrode will be placed on the skin overlying the supraorbital region ipsilateral to the affected area. The current will be delivered at the intensity of 2mA for 20 minutes. To deliver sham, the current will be delivered for 30 sec only to elicit tingling skin sensation but no cortical excitability changes.

SUMMARY:
A study to determine if transcranial direct current stimulation (tDCS, the device that regulates brain activity, can improve pain in people with neuropathic facial pain and compare which modality (inhibitory tDCS over the somatosensory cortex or excitatory tDCS over the motor cortex) can result in better pain-relief.)

DETAILED DESCRIPTION:
This is a pilot study designed to collect preliminary data on safety and efficacy of transcranial direct current stimulation (tDCS)to relieve pain in subjects with neuropathic facial pain,and to compare two pain-treatment tDCS modalities: inhibitory tDCS stimulation over the somatosensory cortex and excitatory tDCS over the motor cortex.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous facial neuropathic pain due to any of following:

  1. Trigeminal neuralgia, type 1, (TN1): facial pain of spontaneous onset with predominantly episodic pain.
  2. Trigeminal neuralgia, type 2, (TN2): facial pain of spontaneous onset with predominantly constant pain.
  3. Trigeminal neuropathic pain, (TNP): facial pain resulting from unintentional injury to the trigeminal system from facial trauma, oral surgery, ear, nose and throat (ENT) surgery, root injury from posterior fossa or skull base surgery, stroke, etc.
  4. Trigeminal deafferentation pain, (TDP): facial pain in a region of trigeminal numbness resulting from intentional injury to the trigeminal system from neurectomy, gangliolysis, rhizotomy, nucleotomy, tractotomy, or other denervating procedures.
  5. Symptomatic trigeminal neuralgia, (STN): facial pain resulting from multiple sclerosis.

  e) Postherpetic neuralgia, (PHN): facial pain resulting from trigeminal Herpes zoster (shingles) outbreak in the trigeminal distribution.
* Pain intensity score for "worst pain in the last 24 hours" >4 on a numeric scale 0-10 at the time of enrollment and before the first stimulation of each treatment block.
* Pain intensity score for "pain right now" >4 on a numeric scale 0-10 before the first stimulation of each block of treatment.

Exclusion Criteria:

* Uncontrolled hypertension, uncontrolled diabetes, uncontrolled cardiovascular disease
* Other painful conditions than neuropathic facial pain, that are not related to and can't be distinguished from the neuropathic facial pain
* Pregnancy
* Implanted neurostimulation devices (e.g. a spinal cord stimulator, a deep brain stimulator, etc)
* Active illegal drug/alcohol abuse
* Unable to follow directions or complete tools in English.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be a composite measure "Pain intensity/consumption of pain medication". | Daily from Baseline to up to 17 weeks
  The washout period between phase I and phase II of the study is variable as patients have to go back to their baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Hao, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States